CLINICAL TRIAL: NCT03160911
Title: The Use of Over-the-scope-clip (OTSC) Versus Standard Therapy for the Prevention of Rebleeding in High Risk Peptic Ulcers: a Randomised Controlled Trial.
Brief Title: The Use of Over-the-scope-clip for Prevention of Rebleeding in High Risk Peptic Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Resident Specialist, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016.711-T
Record Dates: First submitted 2017-05-14; First posted 2017-05-19 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Ulcer Bleeding; Upper Gastrointestinal Tract Bleeding
Keywords: Over-the-scope clip; endoscopic haemostasis

STUDY DESIGN:
Intervention Model Description: There are two separate interventional arms. In case of treatment failure, the two groups are allowed to crossover to the other group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, the investigator and the outcome assessor would be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Over-the-scope clip (Experimental): The patient would receive an esophagogastroduodenoscope to identify the bleeding source. The endoscopist can decided whether to pre inject the ulcer with adrenaline. Then the OTSC is used for haemostasis.
  Interventions: Device: Over-the-scope clip (OTSC)
- Conventional endoscopic haemostasis (Active Comparator): The patient would receive an esophagogastroduodenoscope to identify the bleeding source. Haemostasis will be performed in the conventional way, either using heater probe, endoscopic clips and/or injection of adrenaline
  Interventions: Device: Conventional Endoscopic Haemostasis

INTERVENTIONS:
Device: Over-the-scope clip (OTSC) — The device provides a robust and strong tissue apposition. The system was developed to close perforations and treat bleeding in the gastrointestinal tract. In chronic ulcers, an anchor device can be used to pull the ulcer base toward the aspiration cap to facilitate accurate clip application. Endoscopic haemostasis would be achieved with the use of this device and/or injection of adrenaline
  Arms: Over-the-scope clip
Device: Conventional Endoscopic Haemostasis — This includes the use of heater probe, endoscopic clipping and injection of adrenaline for endoscopic haemostasis
  Arms: Conventional endoscopic haemostasis

SUMMARY:
Non-variceal acute gastrointestinal bleeding is a common and potentially life-threatening problem. The conventional treatment of this condition is for esophagogastroduodenoscopy (OGD) for haemostasis. Treatment methods include heater probe, clipping and injection of adrenaline. Recently, a new device called the Over-the-scope clip (OTSC) has been device to treat perforations and bleeding in the gastrointestinal tract. Therefore, the aim of the study is to compare between the treatment outcomes between OTSC and conventional endoscopic haemostatic methods in ulcers that are of high risk for rebleeding.

DETAILED DESCRIPTION:
Acute upper gastrointestinal bleeding is a common and potentially life-threatening condition. Non-variceal bleeding accounts for more than 80-90% of the cause with gastroduodenal peptic ulcer being the major cause. Endoscopic haemostasis has significantly improved the outcome of these patients. Recurrent bleeding remains one of the most important predictors of mortality. Previous studies have identified ulcers that are high risk for rebleeding.

Conventionally, endoscopic haemostasis is achieved by injection therapy, thermocoagulation or mechanical therapy such as haemostatic clips. However, there are limitations to thermo-coagulation and conventional haemostatic clips. Over the past few years, a novel endoscopic clipping device, the Over-The-Scope Clip (OTSC; Oversco Endoscopy AG, Tübingen, Germany) has become available. The device provides a robust and strong tissue apposition. The system was developed to close perforations and treat bleeding in the gastrointestinal tract. In chronic ulcers, an anchor device can be used to pull the ulcer base toward the aspiration cap to facilitate accurate clip application. With a larger jaw width and greater strength, the OTSC is expected to have superior haemostatic properties when compared to hemo-clips. Case series have been published on the clinical experience of OTSC on gastrointestinal bleeding with promising results.

Therefore, in this randomised controlled trial, we aim to compare the efficacy of the OTSC to standard endoscopic therapy in primary treatment of patients with peptic ulcer bleeding that are of high-risk for rebleeding. The hypothesis is that the use OTSC can significantly decrease the rebleeding rate in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Actively bleeding peptic ulcers (Forrest Ia, Ib), ulcers with non-bleeding visible vessel or Forrest IIa ulcer (defined as protuberant discoloration, or ulcers with an initial clot and upon irrigation shows a vessel) AND
2. Ulcer size ≥ 1.5 cm as determined by an opened biopsy forceps;

Exclusion Criteria:

1. Patients aged below 18
2. Peptic ulcer with concomitant perforation
3. Tumor bleeding
4. Variceal bleeding
5. Patients who are pregnant or lactating
6. Moribund patients or patients with terminal malignancy or end-stage non-malignant conditions, in whom life expectancy is less than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
The number of cases that develop clinical rebleeding | Within 30 days of therapy
  Clinical rebleeding is defined as fresh hematemesis, fresh melena or hematochezia and signs of hypovolemic shock (systolic blood pressure of <90mmHg and pulse rate >110 per minute) and/or a drop in hemoglobin of > 2 g/dl per 24 hours despite adequate transfusion. Rebleeding would be confirmed by an immediate endoscopy showing fresh blood in stomach or active bleeding from a previously seen ulcer. A clinical rebleeding will be independently reviewed by an adjudication panel.

SECONDARY OUTCOMES:
Number of cases that died | within 30 days of therapy
  Death from all causes within 30 days of therapy
Number of units of blood transfusion required in each patient | within 30 days of therapy
  Number of units of blood transfusion required in each patient within 30 days of therapy
Hospital stay | up to one year
  Hospital stay for the episode of bleeding
Number of cases with failure of achieving primary haemostasis | Within 30 days of therapy
  The number of cases with failure of achieving primary haemostasis. Failure of primary haemostasis is defined by the inability to achieve haemostasis during the index endoscopy.
The number of cases requiring further interventions such as repeat endoscopy, surgery or transarterial embolization | Within 30 days of therapy
  The number of cases requiring further interventions such as repeat endoscopy, surgery or transarterial embolization
Hospital costs | Up to one year
  The total direct costs required for the hospital admission for the episode of bleeding measured in Hong Kong dollars

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Chan, MBCHB, FRCS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The IPD will only be used for the purposes of this study and not be disclosed to researchers of outside of this study.

REFERENCES:
- [Derived] Chan S, Pittayanon R, Wang HP, Chen JH, Teoh AY, Kuo YT, Tang RS, Yip HC, Ng SKK, Wong S, Mak JWY, Chan H, Lau L, Lui RN, Wong M, Rerknimitr R, Ng EK, Chiu PWY. Use of over-the-scope clip (OTSC) versus standard therapy for the prevention of rebleeding in large peptic ulcers (size >/=1.5 cm): an open-labelled, multicentre international randomised controlled trial. Gut. 2023 Apr;72(4):638-643. doi: 10.1136/gutjnl-2022-327007. Epub 2022 Oct 28. PMID 36307177